CLINICAL TRIAL: NCT07072533
Title: Effect of Blood Flow Restriction With Aerobic Training on Chest Muscles in Diaplegic Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salah Eid Ahmed Ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SREC.PT.SUE(11)625
Record Dates: First submitted 2025-06-28; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Group A which is the experimental group treated with blood flow restriction plus aerobic training and group B which is the control group treated with aerobic trainin only.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction combined with aerobic training (Experimental): individual will do blood flow restriction aerobic training
  Interventions: Other: blood flow restriction training
- aerobic training only (Active Comparator): individual will do aerobic training
  Interventions: Other: blood flow restriction training

INTERVENTIONS:
Other: blood flow restriction training — individual will do aerobic training .
  Other Names: aerobic training

SUMMARY:
To evaluate the effect of blood flow restriction combined with aerobic training on chest muscle strength in individual with diaplegic cerebral palsy

DETAILED DESCRIPTION:
combining blood flow restriction with aerobic training may enhance muscle function and endurance by increasing localized metabolic stress and systemic cardiovascular effects inducing muscular hypertrophy and strength gaining with low load training especially chest muscles which affected in individuals with diaplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

diaplegic cerebral palsy. GMFCS level I-III. medically stable.

Exclusion Criteria:

severe cognitive impairment. cardio respiratory contraindication. previous thoracic surgery or musculoskeletal deformities affecting chest.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Chest muscle strength | 3 months
  chest muscle strength will be measured by handheld dynamometry measured in Newton

SECONDARY OUTCOMES:
pulmonary function tests | 3 months
  pulmonary function tests in the form of forced vital capacity and forced expiratory volume in one second will be measured in Liters
sub-maximal aerobic capacity | 3 months
  sub-maximal aerobic capacity will be measured using six minute walk test measured in seconds
quality f life | 3 months
  quality f life will be measured using the pediatric quality of life inventory measured in scores from zero point to four points
oxygen saturation and heart rate response | 3 months
  oxygen saturation and heart rate response will be measured using pulse oximeter measured in percentage for oxygen saturation and pulses per minute for heart rate